CLINICAL TRIAL: NCT03928717
Title: A Text-Based Adherence Game for Young People Living With HIV in Ghana
Acronym: TAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Nicholas Tarantino, Sr. Research Scientist, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1227391; K23MH114632 (NIH)
Record Dates: First submitted 2019-04-23; First posted 2019-04-26 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: HIV/AIDS; Medication Adherence
Keywords: adherence; young adult; Africa; mhealth; adolescent; viral load
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text-Based Adherence Game (Experimental): Participants in the experimental condition will receive the Text Based Adherence Game. They will receive semi-automated text messages sent by study staff throughout the trial period.
  Interventions: Behavioral: Text-Based Adherence Game; Behavioral: Standard of Care (SOC)
- Standard of Care (SOC) (Active Comparator): SOC participants will receive the Standard of Care Intervention which includes receiving a brief adherence counseling session and access to clinic resources, including counseling services, throughout the trial period.
  Interventions: Behavioral: Standard of Care (SOC)

INTERVENTIONS:
Behavioral: Text-Based Adherence Game — A mobile health intervention facilitated by a cloud-hosted web application and designed to promote adherence to HIV care through text message-delivered gamification strategies including peer comparison, point reinforcement, feedback on adherence outcomes, facilitation of social support, and use of an engaging and culturally-relevant story-line.
  Arms: Text-Based Adherence Game
Behavioral: Standard of Care (SOC) — A 10- to 20-minute in-person intervention led by a trained HIV treatment adherence counselor focused on providing basic knowledge of HIV and HIV treatment, motivating participants to engage in HIV treatment, and problem-solving barriers to adherence.

SUMMARY:
This study will develop and evaluate a game-based, text message intervention to promote adherence to HIV care among young people living with HIV (YPLH) in Ghana. Intervention development will be guided by feedback from YPLH, their treatment supporters, and clinic staff, consultation with a mobile health services team, and Social Action Theory. Patient participants will be recruited from an urban HIV clinic in Accra, Ghana to complete a randomized pilot of the intervention. All participants will receive a brief adherence counseling session and complete three assessments over the course of 12 months following enrollment. During this time, intervention participants will receive text messages and phone calls from a semi-automated text message system, clinic staff, and other individuals in their life (e.g., family, friends, and partners) who they have identified as supportive of their treatment. The study will provide a wealth of knowledge about YPLH in Ghana, a group vulnerable to poor treatment outcomes, and provide preliminary data on a novel adherence promotion intervention.

DETAILED DESCRIPTION:
Maintaining lifelong adherence to HIV care is a major challenge for older adolescents and young adults (young people) living with HIV in sub-Saharan Africa where HIV infection is globally most prevalent. Innovative, low cost, and easily scaled strategies are urgently needed to improve young people's engagement to HIV treatment and reduce the public health consequences associated with nonadherence including secondary transmission of HIV infection. Modern mobile health (mHealth) interventions improve adherence to care among young people but are currently not feasible for many low-resource areas of sub-Saharan Africa. This includes theory-driven applications that use gamification, where real-life adherence behaviors are combined with interesting story-lines in a mobile game to promote HIV treatment engagement. Whereas web and smartphone access can be limited, traditional cellphones and text messaging are near universal and have been used previously to promote adherence through simple reminders and linkage to staff support in sub-Saharan Africa. However, to date, no text message adherence intervention has been enhanced through the use of gamification. To increase access to this potentially powerful intervention approach, the current study will test a novel mHealth intervention that uses text messages to gamify adherence behavior among YPLH in Ghana. Piloting this intervention will provide information on its feasibility and signs of preliminary efficacy. The ultimate goal following is further evaluation and refinement will be to disseminate the intervention on a large scale across Ghana and other areas of sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

* Living with HIV
* Reads English and speaks English or a local language (e.g., Twi)
* On antiretroviral therapy
* Access to mobile phone throughout study period
* Able to give consent and not impaired by cognitive or medical limitations as per clinical assessment
* Not involved with another HIV prevention or adherence study
* Evidence of a detectable viral load

Exclusion Criteria:

* None

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Tarantino, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Komfo Anokye Teaching Hospital, Kumasi, Ghana

REFERENCES:
- [Derived] Tarantino N, Norman B, Enimil A, Asibey SO, Martyn-Dickens C, O'Neill K, Guthrie KM, Kwara A, Bock B, Mimiaga MJ, Brown LK. Randomized Pilot Trial of the Text-Based Adherence Game for Ghanaian Youth with HIV. AIDS Behav. 2025 Mar;29(3):791-803. doi: 10.1007/s10461-024-04560-3. Epub 2024 Dec 24. PMID 39719465
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Text-Based Adherence Game | Standard of Care (SOC)
Started | 30 | 30
Completed | 25 | 27
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text-Based Adherence Game | Standard of Care (SOC) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.10 (1.94) | 20.57 (2.01) | 20.33 (1.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 16 | 17 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 30 | 60
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Ghana | 30 | 30 | 60
Visual Analog Scale Past 28-Day Adherence [Mean (Standard Deviation); unit: units on a scale] — The is the Visual Analog Scale which measures past 28-day antiretroviral adherence with a single item. Higher scores equal greater adherence. The scale ranges from 0 to 10.
  units on a scale | 6.57 (3.65) | 7.90 (2.81) | 7.23 (3.30)

OUTCOME MEASURES:

1. Primary Outcome: HIV-1 Viral Load (log10 Transformed)
Description: This is a measure of the number of copies of HIV in a person's blood (i.e., copies per ml). It was assessed through blood draw and lab testing. For analyses, raw viral load was log10 transformed to reduce skewness.
Time Frame: Past 90 days
Population: Analyses were conducted with participants who had viral load data at all three time points (n = 48).
Measure: Mean (Standard Deviation); unit: log10 HIV copies/mL
Arm/Group | Text-Based Adherence Game | Standard of Care (SOC)
Number analyzed (Participants) | 23 | 25
log10 HIV copies/mL | 2.22 (1.44) | 2.18 (1.35)
Statistical Analysis 1: Comparison: Text-Based Adherence Game vs Standard of Care (SOC); Test type: Superiority; p < 0.05, ANOVA; Mean Difference (Final Values) = .01

2. Primary Outcome: Self-reported Medication Adherence
Description: The 3-item Self-Report Medication Adherence Scale is used to measure self-reported antiretroviral adherence in the past 30 days. Responses to each of the three items are linearly transformed to a 0-100 scale with zero being the worst adherence and 100 the best. A total score is calculated as the mean of the three individual item scores and ranges from 0 to 100.
Time Frame: Past 30 days
Population: Analyses were conducted with participants who had completed survey assessments at all three time points (n = 51).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Text-Based Adherence Game | Standard of Care (SOC)
Number analyzed (Participants) | 25 | 26
units on a scale | 80.73 (17.32) | 84.03 (15.49)
Statistical Analysis 1: Comparison: Text-Based Adherence Game vs Standard of Care (SOC); Test type: Superiority; p < 0.05, ANOVA; Mean Difference (Final Values) = .16

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Text-Based Adherence Game | Standard of Care (SOC)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT03928717/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT03928717/ICF_001.pdf